CLINICAL TRIAL: NCT07209839
Title: Pelvic Floor Knowledge and Dysfunctions in Female Athletes: Associations With Physical Activity, Demographic Characteristics, and Sports Profile
Brief Title: Pelvic Floor Knowledge and Dysfunction in Female Athletes
Status: Completed | Type: Observational
Sponsor: Berivan Beril Kılıç (Other)
Responsible Party: Sponsor-Investigator, Berivan Beril Kılıç, Assistant Professor, Biruni University
Organization: Biruni University (Other)
Other Study IDs: 4
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Floor; Female Athletes; Physical Activity; Demographic Data
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- female athletes

SUMMARY:
The pelvic floor is a complex structure composed of bones, connective tissue, muscles, and nerves that supports the pelvic organs and provides voluntary control and resting tone of the sphincters. Closely related to continence, sexual function, core stabilization, and posture, the pelvic floor muscles-particularly the levator ani with its type 1 and type 2 fibers-ensure both resting tone and rapid responses to sudden increases in intra-abdominal pressure. In women, pelvic floor dysfunctions (including urinary and anal incontinence, pelvic organ prolapse, defecatory and sexual dysfunctions) occur especially during pregnancy, childbirth, and menopause and adversely affect quality of life. Recently, research on pelvic floor muscles and dysfunctions in female athletes has grown, with competing hypotheses suggesting that these muscles may be strong yet overloaded and weakened due to excessive training. Sports that increase intra-abdominal pressure, such as running, weightlifting, and gymnastics, may stress the pelvic floor and elevate dysfunction risk. Various studies have shown high prevalences of urinary and anal incontinence and pelvic organ prolapse in athletes, alongside generally low pelvic floor awareness. However, few studies have examined the relationship between physical activity level, type, and duration with pelvic floor dysfunction and awareness together. The present study aims to investigate the effects of physical activity, demographic characteristics, and sporting experience on pelvic floor dysfunctions and pelvic floor knowledge in female athletes.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 16-40 years who are literate
* Engaged in any sport, training at least 1 hour per session, at least 3 days per week

Exclusion Criteria:

* Having cooperation problems preventing completion of the questionnaires
* History of neurological disease
* History of urogynecological surgery

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: female athletes who volunteered to participate
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2025-10-03 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Demographic Information Assessment | enrollment
  Participants included in the study will be asked about their age, height, weight, education level, type of sport, years of sporting experience, and history of surgery and illness. They will then be asked to respond to questions, based on a diagram created by the researchers, regarding the location of the pelvic floor, the functions of the pelvic floor muscles, and whether they have experienced pelvic floor-related problems during training. All information will be recorded in the patient tracking form.
Pelvic Floor Health Knowledge Level | enrollment
  Participants' knowledge of pelvic floor health will be assessed using the Pelvic Floor Health Knowledge Test developed by Al-Deges (2019), which aims to measure individuals' knowledge regarding pelvic floor problems. This questionnaire consists of 29 items designed to evaluate knowledge of pelvic floor function and dysfunction. Items 1-8 address pelvic floor function and dysfunction, items 9-21 cover risk factors and etiology, and items 22-29 pertain to diagnosis and treatment. Participants will be asked to answer each item by selecting "yes," "no," or "don't know." The validity and reliability of the questionnaire have been supported by previous studies.
Pelvic Floor Dysfunction | enrollment
  Participants' pelvic floor dysfunctions will be assessed using the Pelvic Floor Distress Inventory-20 (PFDI-20). This scale is designed to evaluate all symptoms related to pelvic floor disorders and the severity of the distress they cause. The PFDI-20 consists of 20 items across three subscales, with responses scored from 0 (not at all) to 4 (quite a bit). Subscale scores are calculated by averaging the responses for each subscale and multiplying by 25, resulting in a score range of 0 to 100 per subscale, and a total score ranging from 0 to 300. The Turkish validity and reliability of the scale were established by Çelenay et al. (2012).
Physical Activity Level | enrollment
  Participants' physical activity levels will be assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). The IPAQ-SF is a widely used, self-reported, valid, and reliable tool designed to determine individuals' physical activity levels over the past seven days. The questionnaire consists of seven items and evaluates walking, moderate, and vigorous physical activities, as well as daily sitting time. It aims to determine the duration and frequency of these activities during the week. Data will be converted into MET (Metabolic Equivalent - MET minutes/week) values for analysis. Based on the total MET score, participants' physical activity levels will be classified as low, moderate, or high. The validity and reliability of the Turkish version of the IPAQ-SF have been established by Sağlam et al. (2010).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Faculy of Medicine-Department of Sports Medicine, Fatih, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Verbeek M, Hayward L. Pelvic Floor Dysfunction And Its Effect On Quality Of Sexual Life. Sex Med Rev. 2019 Oct;7(4):559-564. doi: 10.1016/j.sxmr.2019.05.007. Epub 2019 Jul 24. PMID 31351916
- [Result] Sun C, Hull T, Ozuner G. Risk factors and clinical characteristics of rectal prolapse in young patients. J Visc Surg. 2014 Dec;151(6):425-9. doi: 10.1016/j.jviscsurg.2014.07.013. Epub 2014 Sep 18. PMID 25242503
- [Result] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Result] Magor J, Martin R, Bird ML. Athletes' Knowledge of Pelvic Floor Dysfunction and Their Knowledge of and Engagement with Pelvic Floor Muscle Training: A Scoping Review. Int J Environ Res Public Health. 2025 Jan 14;22(1):104. doi: 10.3390/ijerph22010104. PMID 39857557
- [Result] Machin SE, Mukhopadhyay S. Pelvic organ prolapse: review of the aetiology, presentation, diagnosis and management. Menopause Int. 2011 Dec;17(4):132-6. doi: 10.1258/mi.2011.011108. Epub 2011 Nov 25. PMID 22120945
- [Result] Lakhoo J, Khatri G, Elsayed RF, Chernyak V, Olpin J, Steiner A, Tammisetti VS, Sundaram KM, Arora SS. MRI of the Male Pelvic Floor. Radiographics. 2019 Nov-Dec;39(7):2003-2022. doi: 10.1148/rg.2019190064. PMID 31697623
- [Result] Lai HH, Hsu EI, Teh BS, Butler EB, Boone TB. 13 years of experience with artificial urinary sphincter implantation at Baylor College of Medicine. J Urol. 2007 Mar;177(3):1021-5. doi: 10.1016/j.juro.2006.10.062. PMID 17296403
- [Result] High R, Thai K, Virani H, Kuehl T, Danford J. Prevalence of Pelvic Floor Disorders in Female CrossFit Athletes. Female Pelvic Med Reconstr Surg. 2020 Aug;26(8):498-502. doi: 10.1097/SPV.0000000000000776. PMID 31498240
- [Result] Haylen BT, Maher CF, Barber MD, Camargo S, Dandolu V, Digesu A, Goldman HB, Huser M, Milani AL, Moran PA, Schaer GN, Withagen MI. An International Urogynecological Association (IUGA) / International Continence Society (ICS) joint report on the terminology for female pelvic organ prolapse (POP). Int Urogynecol J. 2016 Feb;27(2):165-94. doi: 10.1007/s00192-015-2932-1. PMID 26755051
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Result] Giagio S, Salvioli S, Pillastrini P, Innocenti T. Sport and pelvic floor dysfunction in male and female athletes: A scoping review. Neurourol Urodyn. 2021 Jan;40(1):55-64. doi: 10.1002/nau.24564. Epub 2020 Nov 2. PMID 33137211
- [Result] Donnelly GM, Moore IS. Sports Medicine and the Pelvic Floor. Curr Sports Med Rep. 2023 Mar 1;22(3):82-90. doi: 10.1249/JSR.0000000000001045. PMID 36866951
- [Result] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Result] Toprak Celenay S, Akbayrak T, Kaya S, Ekici G, Beksac S. Validity and reliability of the Turkish version of the Pelvic Floor Distress Inventory-20. Int Urogynecol J. 2012 Aug;23(8):1123-7. doi: 10.1007/s00192-012-1729-8. Epub 2012 Mar 29. PMID 22456806
- [Result] Casey EK, Temme K. Pelvic floor muscle function and urinary incontinence in the female athlete. Phys Sportsmed. 2017 Nov;45(4):399-407. doi: 10.1080/00913847.2017.1372677. Epub 2017 Sep 5. PMID 28845723
- [Result] Campbell KG, Batt ME, Drummond A. Prevalence of pelvic floor dysfunction in recreational athletes: a cross-sectional survey. Int Urogynecol J. 2023 Oct;34(10):2429-2437. doi: 10.1007/s00192-023-05548-8. Epub 2023 May 10. PMID 37162534
- [Result] Bø, K. Exercise and pelvic floor dysfunction in female elite athletes. Handbook of Sports Medicine and Science: The Female Athlete, 2014, 76-85.
- [Result] Barber MD, Kuchibhatla MN, Pieper CF, Bump RC. Psychometric evaluation of 2 comprehensive condition-specific quality of life instruments for women with pelvic floor disorders. Am J Obstet Gynecol. 2001 Dec;185(6):1388-95. doi: 10.1067/mob.2001.118659. PMID 11744914
- [Result] Aoki Y, Brown HW, Brubaker L, Cornu JN, Daly JO, Cartwright R. Urinary incontinence in women. Nat Rev Dis Primers. 2017 Jul 6;3:17042. doi: 10.1038/nrdp.2017.42. PMID 28681849